CLINICAL TRIAL: NCT04970875
Title: Effect of Parotid Mass Location on Benign Tumor Parotidectomy Scar's Characteristics
Brief Title: Partial Modified Blair Incision on Benign Tumor Parotidectomy Scar's Characteristics
Acronym: MiniBlair
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Ronen Ohad, Director Head and Neck Surgery Unit, Western Galilee Hospital-Nahariya
Other Study IDs: NHR010619
Record Dates: First submitted 2021-06-20; First posted 2021-07-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Salivary Gland Tumor
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — QoL questionnaire

SUMMARY:
Parotidectomy is the treatment of choice for tumors in the parotid gland, with the modified Blair is the most common incision used. In our medical center, the incision is tailored to the size and location of the specific parotid tumor. This retrospective analysis aims to determine the incidence of complications and to assess the relation between the mass and scar characteristics in patients who had undergone parotidectomy.

DETAILED DESCRIPTION:
The scar characteristics of patient who had undergone parotidectomy for benign neoplasms at our medical center between 2013 and 2019 will be evaluated. Patients will complete a questionnaire regarding the occurrence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years during the surgery
* Clinical diagnosis of a benign parotid pathology

Exclusion Criteria:

* A malignant pathology of the parotid gland
* Unavailable data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The scar characteristics of patient who had undergone parotidectomy for benign neoplasms at our medical center between 2013 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by a questionnaire. | 1 Year
  The Warmald Parotidectomy Complications Questionnaire consists of five items, each addressing a complication common to parotidectomy: numbness of the ear on the operated side, Frey's syndrome, facial depression or deformity, noticeable scar, and pain or discomfort in the scar. Subjects are asked to indicate the extent to which they were disturbed by each of these complications on a scale ranging from 1 (never) to 10 (always).

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No